CLINICAL TRIAL: NCT00512772
Title: Improved Use of Antibiotic Guidelines in in Hospital Environment: Research on an Implementation Model and the Role of the Hospital Pharmacist.
Brief Title: Improved Use of Antibiotic Guidelines in Hospital Environment
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Pieter-Jan Cortoos, PharmD, Katholieke Universiteit Leuven
Other Study IDs: B32220072383
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-07

CONDITIONS: Community-Acquired Pneumonia
Keywords: Time series; Implementation
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the use of antibiotic guidelines and thus antibiotics can be improved through a description of possible barriers leading to tailored interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed community-acquired pneumonia (CAP)
* Diagnosed community-acquired pyelonephritis

Exclusion Criteria:

* CAP: hospital-acquired pneumonia; patients transferred from other hospital; death within 24h, aspiration pneumonia, immunocompromised status, palliative status, admission due to social reasons
* Pyelonephritis: urinary tract with functional or physical abnormalities, urinary catheterisation, pregnancy, (immunocompromised status, palliative status, admission due to social reasons and history of renal transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with a diagnosis of community-acquired pneumonia or community-acquired pyelonephritis
Sampling Method: Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter-Jan Cortoos, PharmD, Principal Investigator — KU Leuven; Gert Laekeman, PhD, Study Director — KU Leuven
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Gasthuisberg, Leuven